CLINICAL TRIAL: NCT00618436
Title: Assessment of Seizure Prophylaxis Protocols Using Intravenous Levetiracetam in a Neuroscience Intensive Care Unit
Brief Title: Assess Safety and Efficacy of Levetiracetam(LEV;Keppra)for Seizure Prevention
Acronym: Keppra
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Mayfield Clinic & Spine Institute (Other)
Responsible Party: Principal Investigator, Lori Shutter, Director, Neurocritical Care Fellowship Program, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-4-6-7
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
Keywords: Seizures; Traumatic Brain Injury; Subarachnoid Hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Seizures | interventions — Levetiracetam; Phenytoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Active Comparator): Group 1 - The levetiracetam (Keppra®) group will receive a loading dose of 20 mg/kg IV over 15 minutes (rounded to the nearest 250mg) up to a maximum of 2000 mg, then started on maintenance dose (1000 mg, IV BID)as prophylaxis for 7 days.
  Interventions: Drug: Levetiracetam
- Phenytoin (Active Comparator): Group 2-The phenytoin group will receive a loading dose of 20 mg/kg IV to a maximum of 2000mg, then started on maintenance dose at 5 mg/kg/day (rounded to nearest 100mg dose, IV, divided into three doses a day) as prophylaxis for 7 days. Phenytoin levels are to be checked daily and dose adjusted as needed to maintain therapeutic levels of 10-20 µg/dL.
  Interventions: Drug: Phenytoin

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam group will receive a loading dose of 20 mg/kg IV(rounded to nearest 250mg) to a maximum of 2000mg, then started on maintenance dose (1000 mg,IV q 12h) as prophylaxis for seven days.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Phenytoin — The group will receive a loading dose of fosphenytoin 20 mg/kg IV to a maximum of 2000 mg, then started on maintenance dose of 5mg/kg/day, rounded to nearest 100mg dose, IV, q 12h for seven days.
  Other Names: Dilantin
  Arms: Phenytoin

SUMMARY:
To show that the use of intravenous levetiracetam(LEV;Keppra)for seizure prevention in patients in the Neuroscience Intensive Care Unit will result in fewer side effects compared to the current standard of care anticonvulsant and will be at least as effective as the current standard of care in preventing clinical and sub-clinical seizure activity.

DETAILED DESCRIPTION:
To show that the use of intravenous levetiracetam(LEV;Keppra)for seizure prophylaxis in the Neuroscience Intensive Care Unit will result in fewer adverse effects compared to the current standard of care anticonvulsant(phenytoin) and will be at least as effective as phenytoin in preventing clinical and sub-clinical seizure activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with traumatic brain injury
* Glasgow Coma Score (GCS) score 3-8(inclusive),or GCS motor score of 5 or less and abnormal admission CT scan showing intracranial pathology
* Hemodynamically stable with a systolic BP >90 mm Hg
* At least one reactive pupil
* A negative pregnancy test in females
* Age at least 18 years
* Signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for research form OR
* Subjects with subarachnoid hemorrhage (SAH)
* SAH documented by CT scan
* Hunt-Hess grade 3-5, inclusive
* Hemodynamically stable with a systolic BP> 90 mm Hg
* At least one reactive pupil
* A negative pregnancy test in females
* Age of at least 18 years
* Signed informed consent and HIPAA authorization for research form

Exclusion Criteria for enrollment

* No venous access
* Spinal cord injury
* History of or CT confirmation of previous brain injury such as brain tumor, cerebral infarct, or spontaneous intracerebral hemorrhage
* Hemodynamically unstable
* Suspected anoxic events
* Other peripheral trauma likely to result in liver failure
* Positive pregnancy test in females
* Age less than 18 years of age
* Known hypersensitivity to any anticonvulsant
* An injury that, in the opinion of the principal investigator, has a high likelihood of death within the first 72 hours.
* Any treatment, condition, or injury that contraindicates treatment with LEV (levetiracetam) or phenytoin (PHT).
* Inability to obtain signed informed consent or HIPAA authorization for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Shutter, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Cincinnati Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Steinbaugh LA, Lindsell CJ, Shutter LA, Szaflarski JP. Initial EEG predicts outcomes in a trial of levetiracetam vs. fosphenytoin for seizure prevention. Epilepsy Behav. 2012 Mar;23(3):280-4. doi: 10.1016/j.yebeh.2011.12.005. Epub 2012 Feb 16. PMID 22342434

RESULTS

PARTICIPANT FLOW:
Groups:
- Levetiracetam: This group will receive treatment with Levetiracetam.
- Phenytoin: This group will receive treatment with Phenytoin.
Period: Overall Study
Arm/Group | Levetiracetam | Phenytoin
Started | 34 | 18
Completed | 34 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient was enrolled at 17 years of age. His age was unknown at the time of admission to the hospital after his trauma, and based on body size/habitus he appeared to be a young adult. It was later discovered that he was only 17, but turning 18 in 3 days. The PI decided to allow his participation in the study at the parents request.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Phenytoin | Total
Number analyzed (Participants) | 34 | 18 | 52
Age, Continuous [Median (Full Range); unit: years] | 44 [17 to 75] | 35 [18 to 80] | 42.5 [17 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 26 | 13 | 39
Region of Enrollment [Number; unit: participants]
  United States | 34 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Seizure Incidence
Description: This was the number of patients in each group who demonstrated seizure activity during the course of the study
Time Frame: Duration of study, up to 6 months after the injury
Measure: Number; unit: Participants
Arm/Group | Levetiracetam | Phenytoin
Number analyzed (Participants) | 34 | 18
Participants | 5 | 3

2. Secondary Outcome: Extended Glasgow Outcome Score
Description: This is an 8 point validated scale that measures disability after brain injury. It is assessed through an in person exam or by phone interview at hospital discharge, 3 months and 6 months after injury. The categories are: 1 = dead; 2 = vegetative state; 3 = severe disability, low level; 4 = severe disability, high level; 5 = moderate disability, low level; 6 = moderate disability, high level; 7 = good recovery - low level; 8 = good recovery - high level. Specific questions and activities are assessed to determine into which category the patient falls.
Time Frame: at discharge; 3 and 6 months following injury
Population: All patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Levetiracetam | Phenytoin
Number analyzed (Participants) | 34 | 18
units on a scale
  At Discharge | 2 [1 to 4] | 2 [1 to 3]
  At 3 months | 3 [1 to 7] | 3 [1 to 5]
  At 6 months | 3 [1 to 8] | 3 [1 to 7]

3. Secondary Outcome: Disability Rating Scale (DRS)
Description: The Disability rating scale (DRS) is frequently used in the rehabilitation literature as a measure of disability. It is a reliable, easily performed test that assesses 8 items (eye opening, verbalization, motor response, feeding, toileting, grooming, level of functioning, employability), and assigns each a numerical score ranging from 0 - 5 based on the category. The domains these 8 items are felt to assess include: alertness, cognition for self-care, dependence, and psychosocial adaptability. The scoring range is from 0-30, with increasing disability levels assigned to higher numerical values. The total DRS is then dichotomized into favorable (disability = none, mild, partial or moderate disability) and unfavorable (disability = moderately severe, severe, extremely severe, vegetative state, extreme vegetative state, death) outcomes. A DRS score of 0-6 was favorable, with any score greater than 6 categorized as unfavorable.
Time Frame: Discharge; 3 and 6 months following injury
Population: All patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Levetiracetam | Phenytoin
Number analyzed (Participants) | 34 | 18
units on a scale
  At Discharge | 24 [7 to 30] | 23 [7 to 30]
  At 3 months | 15 [0 to 30] | 13 [5 to 30]
  At 6 months | 17 [0 to 30] | 9 [0 to 30]

4. Secondary Outcome: Incidence of Adverse Events
Time Frame: discharge; 3 and 6 months following injury
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Levetiracetam | Phenytoin
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/18
Other Adverse Events (participants affected / at risk) | 0/34 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No